CLINICAL TRIAL: NCT06231381
Title: A Phase II, Multicenter, Double-blind, Randomized, Placebo Parallel-controlled Trial to Evaluate the Efficacy and Safety of HB0034 in Patients with GPP Presenting with an Acute Flare of Moderate to Severe Intensity
Brief Title: Efficacy and Safety of HB0034 in Patients with Generalized Pustular Psoriasis (GPP)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Huaota Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HB0034-04
Record Dates: First submitted 2024-01-21; First posted 2024-01-30 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Generalized Pustular Psoriasis (GPP)
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HB0034 (Active Comparator): Subjects will be given a single intravenous infusion of HB0034 on D1.
  Interventions: Drug: HB0034
- Placebo (Placebo Comparator): Subjects will be given a single intravenous infusion of placebo on D1.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: HB0034 — Anti-IL-36R antibody
  Other Names: Recombinant Humanized anti-IL-36R Monoclonal antibody
  Arms: HB0034
Other: Placebo — non-biologically active drug
  Arms: Placebo

SUMMARY:
This is a phase II, multicenter, double-blind, randomized, placebo parallel-controlled clinical trial to evaluate the efficacy and safety of HB0034 in patients with generalized pustular psoriasis (GPP) presenting with an acute flare of moderate to severe intensity.

DETAILED DESCRIPTION:
GPP patients who are experiencing an acute flare will be screened. Before randomization, the investigator must ensure that the subjects meet all inclusion criteria and do not meet any exclusion criteria.

Subjects will be given a single intravenous infusion of HB0034 or placebo (2:1) on D1 and be hospitalized for at least 8 days after administration of the study drug (including Day 1 for administration). Thereafter, the decision of the patient's discharge will be left at the discretion of the investigator and based on the evolution of the GPP flare and the patient's health status.

Subjects will be followed up to W12-W20.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be experiencing an acute GPP flare of moderate-to-severe intensity at baseline, defined as:

  1. A Generalized Pustular Psoriasis Physician Global Assessment (GPPGA) score of ≥ 3;
  2. New appearance or worsening of existing pustules, and a GPPGA pustulation subscore of ≥ 2;
  3. ≥ 5% Body Surface Area (BSA) covered with pustules.
* Men and women of reproductive age who have no parenting plans and are willing to use reliable contraception during the study period and for 6 months after the last dose of the study drug;
* Patients who fully understand and voluntarily sign an ICF, and are willing and able to follow clinical study and subsequent visit schedules.

Exclusion Criteria:

* Drug-triggered acute generalized exanthematous pustulosis (AGEP);
* Synovitis-acne-pustulosis-hyperostosis-osteitis syndrome (SAPHO);
* Other active inflammatory or autoimmune diseases requiring systemic treatment with immunosuppressants, including but not limited to rheumatoid arthritis (RA), psoriatic arthritis (PsA), systemic lupus erythematosus (SLE), inflammatory bowel disease, and uveitis.
* Patients with an increased risk of infectious complications as assessed by the investigator (e.g., a recent suppurative infection, any congenital or acquired immunodeficiency, such as HIV infection, prior organ or stem cell transplantation);
* Patients who have received a live vaccine or investigational live vaccine within 6 weeks prior to the first dose of the study drug, or plan to receive a live vaccine or participate in a clinical study of investigational live vaccine during the study period or within 6 weeks after completion of administration of the study drug;
* Patients who have had a serious trauma or undergone a major surgery within 1 month prior to the first dose of the study drug, or plan to undergo any elective surgery during the study period;
* Patients with documented active or suspected malignancy or a history of malignancy within 5 years prior to screening;
* Patients with a history of severe allergy, who have experienced grade 3-4 allergic reactions when receiving other monoclonal antibodies, or those who are known to have hypersensitivity to protein drugs, recombinant proteins, or HB0034 components;
* Subjects who are pregnant or breastfeeding, or those who have a positive pregnancy test result. Breastfeeding female subjects who stop breastfeeding prior to the first dose of the study drug until 16 weeks after the end of the trial will not be excluded;
* Patients who are currently participating in clinical trials or have participated in clinical trials of any drug/device within 30 days (or 5 half-lives, whichever is longer) prior to the first dose of the study drug;
* Patients expected to have poor compliance, such as those who are uncooperative, fail to receive follow-up on time, and are unlikely to complete the study;
* Other reasons that the investigator considers it is inappropriate to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who achieved GPPGA pustulation subscore of 0/1 (no/almost no visiable pustules) at Week 1. | Week 1
  Generalized Pustular Psoriasis Physician Global Assessment (GPPGA)

SECONDARY OUTCOMES:
Percent (%) improvement from baseline in GPPASI at Week 1 | Week 1
  Generalized Pustular Psoriasis Area and Severity Index (GPPASI)
Safety endpoints include the proportion of subjects with TEAEs. | 12-20 Weeks
  The safety assessment includes monitoring for AEs, SAEs (including SAEs related to protocol procedures from signing of ICF until before the first dose of the study drug) from the first dose of the study drug to end of study (EOS) , as well as changes from baseline in laboratory tests, vital signs, physical examination, and 12-lead electrocardiogram (ECG).

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking University People's Hospital (PKUPH), Beijing
  - Shanghai Huaota Biopharmaceutical Co., Ltd, Shanghai

IPD SHARING:
Plan to Share IPD: No